CLINICAL TRIAL: NCT00120939
Title: Phase I Trial of Motexafin Gadolinium (MGd) and Docetaxel Chemotherapy in the Treatment of Advanced Solid Tumors
Brief Title: Study of Motexafin Gadolinium and Docetaxel for Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0212
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2007-05

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms
Keywords: Lung Cancer; Breast Cancer; Prostate Cancer; Ovarian Cancer; Head and Neck Cancer; Gastrointestinal Cancer; Metastatic Cancer; Advanced Cancer; Genitourinary Cancer; Glioblastoma Multiforme; Recurrent Cancer; Colon Cancer; Gastric Cancer; Stomach Cancer; Pancreatic Cancer; Esophageal Cancer; Throat Cancer; Bladder Cancer; Kidney Cancer; Renal Cancer; Cervical Cancer; Endometrial Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis; Urogenital Neoplasms; Glioblastoma; Recurrence; Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium

SUMMARY:
The primary purpose of this study is to evaluate the safety, side effects, and dosage for Motexafin Gadolinium given with the chemotherapy drug docetaxel to patients with advanced cancers. Secondly, tumor response to the combined treatment, drug levels in the body, and drug interactions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Metastatic, or unresectable solid tumors from breast, head, and neck, gastrointestinal, genitourinary, lung, or ovarian cancer or recurrent glioblastoma multiforme
* ECOG performance status score either 0, 1, or 2
* Willing and able to provide written informed consent

Exclusion Criteria:

* Greater than two prior cytotoxic regimens
* Laboratory values showing adequate function of bone marrow, liver, and kidneys
* Uncontrolled hypertension
* Known sensitivity to or intolerable adverse effects from taxanes (eg. paclitaxel, docetaxel) or polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25

PRIMARY OUTCOMES:
Determine the Dose Limiting Toxicity at 8 weeks (2 cycles), and the Maximum Tolerated Dose at 24 weeks.

SECONDARY OUTCOMES:
Tumor response rate 8, 16 and 24 weeks, and common PK parameters at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal Chatta, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States